CLINICAL TRIAL: NCT00259272
Title: Phase IIIb, Multicenter, Single-Arm Open-Label Study, Supporting the Development and the Validation of the MATHYS Scale (Multidimensional Assessment of THYmic States) in a Population of Bipolar Patients Treated With Olanzapine, Either in-Label (Manic and Mixed Patients) and Off-Label (Hypomanic and Bipolar Depression)
Brief Title: Validation of Multidimensional Assessment of THYmic States (MATHYS): A Study in a Population of Bipolar Patients Treated With Olanzapine
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Chief Medical Officer, Eli Lilly
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 9675; F1D-FP-S057
Record Dates: First submitted 2005-11-28; First posted 2005-11-29 (Estimated); Results first posted 2009-06-24 (Estimated); Last update posted 2009-06-24 (Estimated); Status verified 2009-04

CONDITIONS: Bipolar Disorder I or II
MeSH Terms: interventions — Olanzapine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- A (Experimental)
  Interventions: Drug: olanzapine

INTERVENTIONS:
Drug: olanzapine — 5 to 20 mg (flexible dose) administered orally as disintegrated tablets, daily for 24 weeks.
  Other Names: LY170053; Velotab; Zydis

SUMMARY:
A non randomized study to validate the MATHYS Scale in a population of in and outpatients greater than or equal to 18 years of age, suffering from Bipolar Disorder I or II, and treated with olanzapine.

ELIGIBILITY:
Inclusion Criteria:

1. Patients must meet Diagnostic and Statistical Manual of Mental Disorders, Fourth Edition, Text Revision (DSM-IV-TR) disease diagnostic criteria for Bipolar Disorder

   * currently or most recently in a Manic Episode (Single Manic Episode or Most Recent Episode Manic) or
   * currently or most recently in a Hypomanic Episode or
   * currently or most recently in a Mixed Episode or
   * currently or most recently in a Major Depressive Episode
   * and confirmed by the module D of the SCID (Semi-Structured Interview).
2. Patients must be more than 18 of age at Visit 0.

Exclusion Criteria:

1. A valid current or lifetime DSM-IV-TR Axis I or II diagnosis which could interfere, at the investigator's opinion, with the evaluation.
2. Patients on antidepressant or mood stabilizer therapy one week (four weeks with fluoxetine) prior to Visit 1, with the exception of mood stabilizer therapy considered in the opinion of the investigator as an efficient treatment for at least one year prior to the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 141 (Actual)
Dates: Start 2005-11; Primary Completion 2008-05 (Actual); Study Completion 2008-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon-Fri 9 AM - 5 PM Eastern time (UTC/GMT-5 hours, EST), Study Director — Eli Lilly and Company
Locations (16):
- France (16):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Andilly
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Bordeaux
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Cornebarrieu
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Créteil
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., La Rochelle
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., La Seyne-sur-Mer
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Lyon
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Marseille
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Montpellier
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Nîmes
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Orvault
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Paris
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Pin-Balma
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Plaisir
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Poitiers
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Toulouse

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: All participants received olanzapine and were grouped according to their most recent type of episode.
Groups:
- Manic Episode; Mixed Episode: olanzapine: 5 to 20 mg (flexible dose) administered orally as disintegrated tablets, daily for 24 weeks (initial dose = 15 mg).
- Hypomanic Episode: olanzapine: 5 to 20 mg (flexible dose) administered orally as disintegrated tablets, daily for 24 weeks (initial dose = 10 mg)
- Depressive Episode: olanzapine: 5 to 20 mg (flexible dose) administered orally as disintegrated tablets, daily for 24 weeks (initial dose = 5 mg).
Period: Overall Study
Arm/Group | Manic Episode | Hypomanic Episode | Mixed Episode | Depressive Episode
Started | 36 | 31 | 26 | 48
Completed | 21 | 24 | 21 | 27
Not Completed | 15 | 7 | 5 | 21
Not completed — Adverse Event | 2 | 1 | 0 | 3
Not completed — Lack of Efficacy | 5 | 1 | 2 | 6
Not completed — Physician Decision | 1 | 2 | 1 | 3
Not completed — Protocol Violation | 2 | 0 | 0 | 1
Not completed — Sponsor Decision | 0 | 1 | 0 | 0
Not completed — Withdrawal by Subject | 4 | 2 | 2 | 7
Not completed — Lost to Follow-up | 1 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Manic Episode | Hypomanic Episode | Mixed Episode | Depressive Episode | Total
Number analyzed (Participants) | 36 | 31 | 26 | 48 | 141
Age Continuous [Mean (Standard Deviation); unit: years] | 46.39 (15.32) | 45.81 (11.68) | 46.62 (12.87) | 44.35 (11.98) | 45.61 (12.91)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19 | 21 | 15 | 25 | 80
  Male | 17 | 10 | 11 | 23 | 61
Region of Enrollment [Number; unit: participants]
  France | 36 | 31 | 26 | 48 | 141
Diagnostic Summary [Number; unit: participants]
  Bipolar Disorder I | 36 | 14 | 26 | 31 | 107
  Bipolar Disorder II - Hypomanic | 0 | 17 | 1 | 0 | 18
  Bipolar Disorder II - Depressed | 0 | 0 | 1 | 17 | 18
Number of Lifetime Suicide Attempts [Number; unit: participants]
  Missing Data | 2 | 3 | 1 | 2 | 8
  0 | 24 | 23 | 15 | 28 | 90
  1 | 8 | 3 | 6 | 5 | 22
  2 | 2 | 0 | 3 | 8 | 13
  4 | 0 | 1 | 0 | 2 | 3
  5 | 0 | 0 | 0 | 2 | 2
  6 | 0 | 1 | 0 | 0 | 1
  10 | 0 | 0 | 1 | 1 | 2
Participants with at Least One Episode of Depression [Number; unit: participants] — Presence of at least one previous episode was defined as: number of episodes in the past 12 months reported and/or number of episodes lifetime reported and/or year of onset of the first symptoms reported.
  participants
    Missing Data | 0 | 0 | 1 | 0 | 1
    No | 6 | 2 | 4 | 0 | 12
    Yes | 30 | 29 | 21 | 48 | 128
Participants with at Least One Episode of Hypomania [Number; unit: participants] — Presence of at least one previous episode was defined as: number of episodes in the past 12 months reported and/or number of episodes lifetime reported and/or year of onset of the first symptoms reported.
  participants
    Missing Data | 2 | 0 | 3 | 1 | 6
    No | 30 | 1 | 14 | 25 | 70
    Yes | 4 | 30 | 9 | 22 | 65
Participants with at Least One Episode of Mania [Number; unit: participants] — Presence of at least one previous episode was defined as: number of episodes in the past 12 months reported and/or number of episodes lifetime reported and/or year of onset of the first symptoms reported.
  participants
    Missing Data | 0 | 3 | 1 | 0 | 4
    No | 0 | 14 | 11 | 23 | 48
    Yes | 36 | 14 | 14 | 25 | 89
Participants with at Least One Episode of Mixed Episode [Number; unit: participants] — Presence of at least one previous episode was defined as: number of episodes in the past 12 months reported and/or number of episodes lifetime reported and/or year of onset of the first symptoms reported.
  participants
    Missing Data | 1 | 3 | 1 | 2 | 7
    No | 27 | 25 | 3 | 32 | 87
    Yes | 8 | 3 | 22 | 14 | 47
Patient Status [Number; unit: participants]
  Inpatient | 26 | 12 | 10 | 24 | 72
  Outpatient | 10 | 19 | 16 | 24 | 69
Previous Central Nervous System Treatment [Number; unit: participants]
  Yes | 34 | 30 | 26 | 46 | 136
  No | 2 | 1 | 0 | 2 | 5
Suicide Ideation [Number; unit: participants] — Assessed via the 17-item Hamilton Depression Rating Scale (HAMD-17) item 3. Item 3 assesses presence and level of suicidal ideations.
  participants
    0: Absent | 35 | 29 | 15 | 26 | 105
    1: Feels Life Not Worth Living | 0 | 2 | 8 | 12 | 22
    2:Wishes He Were Dead or Thoughts of Death to Self | 1 | 0 | 3 | 10 | 14
    3: Suicide Ideas or Gestures | 0 | 0 | 0 | 0 | 0
    4: Attempts Suicide | 0 | 0 | 0 | 0 | 0
Thymic Reactivity - Investigator-Based Assessment [Number; unit: participants] — Investigators were asked - according to your clinical experience, is the patient with: neither; thymic hyper-reactivity; or thymic hypo-reactivity.
  participants
    Neither | 1 | 2 | 4 | 3 | 10
    Thymic Hyper-Reactivity | 34 | 28 | 20 | 19 | 101
    Thymic Hypo-Reactivity | 1 | 1 | 2 | 26 | 30
Age at Time of Onset of First Episode [Mean (Standard Deviation); unit: years] | 30.57 (13.94) | 34.00 (13.75) | 27.36 (10.78) | 29.19 (10.41) | 30.29 (12.31)
Body Mass Index [Mean (Standard Deviation); unit: kilogram per meter squared] — Body mass index is an estimate of body fat based on body weight divided by height squared.
  kilogram per meter squared | 24.80 (4.53) | 24.73 (4.98) | 26.86 (7.75) | 24.54 (3.70) | 25.09 (5.18)
Duration of Current Episode [Mean (Standard Deviation); unit: months] | 0.99 (1.51) | 1.95 (3.22) | 1.71 (1.56) | 1.51 (1.49) | 1.53 (2.03)
Duration of Illness [Mean (Standard Deviation); unit: years] | 16.86 (13.93) | 12.45 (9.52) | 19.28 (14.54) | 15.70 (11.59) | 15.91 (12.46)
Weight [Mean (Standard Deviation); unit: kilograms] | 68.83 (12.34) | 69.89 (14.71) | 74.42 (20.00) | 70.85 (14.41) | 70.78 (15.15)

OUTCOME MEASURES:

1. Primary Outcome: Mean Changes From Baseline to 6 Week and 24 Week Endpoints in the Multidimensional Assessment of THYmic States Scale (MATHYS) Total Score
Description: A visual analogic scale consisting of 20 items. Item scores vary from 0 (inhibition of the state evaluated by the item) to 10 (excitation for the evaluated state), except for items 5 to 10 and 17 and 18 which are inversed and are consequently to be reversed before the analysis. Total score is sum of the 20 items and can vary from 0 to 200.
Time Frame: Baseline, 6 Weeks, 24 weeks
Population: Intention to treat. Number of participants with baseline and at least one non-missing postbaseline value.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Manic Episode | Hypomanic Episode | Mixed Episode | Depressive Episode
Number analyzed (Participants) | 36 | 31 | 26 | 48
units on a scale
  Baseline (n=34, 31, 25, 48) | 140.55 (22.18) | 136.52 (22.45) | 116.74 (21.30) | 76.88 (22.91)
  6 Week Endpoint (n=31, 31, 25, 44) | 115.37 (23.09) | 105.15 (23.10) | 101.58 (22.55) | 93.41 (23.71)
  Change from 6 Week Endpoint (n=30, 31, 24, 44) | -22.91 (28.70) | -31.37 (30.46) | -13.32 (26.37) | 17.17 (26.62)
  24 Week Endpoint (n=35, 31, 26, 47) | 115.15 (24.84) | 103.16 (23.03) | 91.56 (25.19) | 94.58 (27.09)
  Change from 24 Week Endpoint (n=34, 31, 25, 47) | -24.67 (24.83) | -33.36 (33.61) | -26.08 (40.51) | 17.04 (31.81)

2. Secondary Outcome: Mean Change From Baseline to 6 Week and 24 Week Endpoints in the Hamilton 17-Items Depression Scale (HAMD-17) Total Score
Description: The 17-item HAMD measures depression severity. Each item was evaluated and scored using either a 5-point scale (e.g. absent, mild, moderate, severe, very severe) or a 3-point scale (e.g. absent, mild, marked). The total score of HAMD-17 may range from 0 (not at all depressed) to 52 (severely depressed).
Time Frame: Baseline, 6 Weeks, 24 Weeks
Population: Intention to treat. Number of participants with baseline and at least one non-missing postbaseline value.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Manic Episode | Hypomanic Episode | Mixed Episode | Depressive Episode
Number analyzed (Participants) | 36 | 31 | 26 | 48
units on a scale
  Baseline (n=35, 30, 26, 48) | 6.46 (4.86) | 8.43 (5.33) | 12.65 (4.83) | 16.06 (7.19)
  Change from 6 Week Endpoint (n=29, 29, 25, 45) | -1.79 (4.59) | -3.10 (4.59) | -5.60 (6.60) | -8.51 (6.22)
  Change from 24 Week Endpoint (n=34, 30, 26, 47) | -1.74 (5.02) | -3.20 (6.40) | -5.50 (6.72) | -7.96 (7.18)

3. Secondary Outcome: Mean Change From Baseline to 6 Week and 24 Week Endpoints in the Hamilton Anxiety Scale (HAMA) Total Score
Description: The 14-item HAMA assesses the severity of anxiety. The investigator talked to the patient about their symptoms over the previous week before the study visit. Each item was scored using a 5-point scale, i.e. 0 = absent to 4 = severe. The total score of HAMA-14 may range from 0 (not present) to 56 (very severe).
Time Frame: Baseline, 6 Weeks, 24 Weeks
Population: Intention to treat. Number of participants with baseline and at least one non-missing postbaseline value.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Manic Episode | Hypomanic Episode | Mixed Episode | Depressive Episode
Number analyzed (Participants) | 36 | 31 | 26 | 48
units on a scale
  Baseline (n=36, 31, 26, 48) | 7.78 (6.29) | 11.94 (7.73) | 15.46 (7.17) | 15.08 (7.35)
  Change from 6 Week Endpoint (n=31, 31, 25, 45) | -2.68 (4.85) | -5.48 (5.89) | -7.32 (6.31) | -6.76 (6.61)
  Change from 24 Week Endpoint (n=35, 31, 26, 47) | -2.26 (4.80) | -5.65 (7.36) | -7.62 (7.87) | -6.83 (7.19)

4. Secondary Outcome: Mean Change From Baseline to 6 Week and 24 Week Endpoints in the Young Mania Rating Scale (YMRS) Total Score
Description: The YMRS is an 11-item scale that measures the severity of manic episodes. Four items are rated on a scale from 0 (symptom not present) to 8 (symptom extremely severe). The remaining items are rated on a scale from 0 (symptom not present) to 4 (symptom extremely severe). The YMRS total score ranges from 0 to 60.
Time Frame: Baseline, 6 Weeks, 24 Weeks
Population: Intention to treat. Number of participants with baseline and at least one non-missing postbaseline value.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Manic Episode | Hypomanic Episode | Mixed Episode | Depressive Episode
Number analyzed (Participants) | 36 | 31 | 26 | 48
units on a scale
  Baseline (n=36, 31, 25, 46) | 24.50 (10.34) | 17.84 (4.88) | 12.96 (7.69) | 2.78 (3.64)
  Change from 6 Week Endpoint (n=31, 31, 24, 43) | -13.65 (9.38) | -13.13 (6.02) | -9.67 (7.91) | -0.86 (3.54)
  Change from 24 Week Endpoint (n=35, 31, 25, 45) | -14.00 (10.94) | -14.45 (7.36) | -10.60 (7.95) | -0.82 (3.24)

5. Secondary Outcome: Mean Change From Baseline to 24 Week Endpoint in Glycaemia Levels (Glucose Fasting Levels)
Time Frame: baseline and 24 weeks
Population: Safety Population. All participants having been prescribed at least one dose of study drug. Number of participants with baseline and at least one non-missing postbaseline value.
Measure: Mean (Standard Deviation); unit: milligrams per deciliter
Arm/Group | Manic Episode | Hypomanic Episode | Mixed Episode | Depressive Episode
Number analyzed (Participants) | 36 | 31 | 26 | 48
milligrams per deciliter
  Baseline (n=33, 30, 23, 47) | 89.27 (16.31) | 85.99 (11.33) | 85.94 (12.58) | 88.52 (13.95)
  Change from 24 Week Endpoint (n=26, 28, 23, 40) | -3.07 (16.15) | 4.65 (15.32) | 3.89 (9.62) | 7.31 (30.42)

6. Secondary Outcome: Increases and Decreases in Fasting Glucose Levels
Time Frame: over 24 weeks
Population: Safety Population. All participants having been prescribed at least one dose of study drug.
Measure: Number; unit: participants
Arm/Group | Manic Episode | Hypomanic Episode | Mixed Episode | Depressive Episode
Number analyzed (Participants) | 36 | 31 | 26 | 48
participants
  At Least One Increase in Fasting Glucose (FG) | 5 | 9 | 3 | 10
  At Least One Decrease in FG | 4 | 8 | 1 | 11
  At Least One Increase/Decrease in FG | 7 | 10 | 3 | 15
  Patients Who Increase and Decrease During Study | 2 | 7 | 1 | 6

7. Secondary Outcome: Mean Change From Baseline to 24 Week Endpoint in Lipids
Description: Baseline, change from baseline, and percent change for the following lipids are presented: Total Cholesterol (TC), High Density Lipoproteins (HDL), Low Density Lipoproteins (LDL), and Triglycerides (TG).
Time Frame: Baseline and 24 Weeks
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: milligrams per deciliter
Arm/Group | Manic Episode | Hypomanic Episode | Mixed Episode | Depressive Episode
Number analyzed (Participants) | 36 | 31 | 26 | 48
milligrams per deciliter
  TC Baseline (n=33, 30, 24, 46) | 182.88 (41.88) | 191.55 (42.49) | 210.51 (50.78) | 203.77 (44.66)
  Change in TC from 24 Week Endpoint (n=26,28,23,41) | 23.64 (33.95) | 2.26 (27.25) | 7.03 (30.77) | 4.41 (50.69)
  Percent Change in TC (n=26, 28, 23, 41) | 14.96 (19.57) | 3.10 (13.83) | 4.41 (16.97) | 4.68 (23.67)
  HDL Baseline (n=33, 30, 23, 46) | 50.21 (14.65) | 56.87 (16.77) | 57.46 (19.13) | 50.78 (13.35)
  Change in HDL from Endpoint (n=26, 28, 22, 41) | 1.24 (13.32) | 1.57 (13.14) | -0.45 (16.27) | 3.25 (12.72)
  Percent Change in HDL (n=26, 28, 22, 41) | 6.04 (26.43) | 6.17 (26.06) | 3.78 (26.12) | 8.87 (23.97)
  LDL Baseline (n=34, 30, 23, 46) | 112.76 (39.81) | 112.16 (31.37) | 129.70 (44.64) | 128.81 (39.26)
  Change in LDL from Endpoint (n=27, 27, 22, 41) | 14.22 (41.05) | 1.28 (36.64) | 9.46 (32.04) | -1.19 (42.24)
  Percent Change in LDL (n=27, 27, 22, 41) | 20.54 (33.94) | 5.15 (33.05) | 11.37 (28.57) | 3.41 (32.28)
  TG Baseline (n=35, 30, 23, 46) | 115.81 (43.15) | 110.66 (89.64) | 131.37 (71.65) | 120.15 (66.63)
  Change in TG from 24 Week Endpoint (n=27,28,22,41) | 8.37 (66.50) | 25.86 (90.32) | -1.16 (49.06) | 13.85 (67.59)
  Percent Change in TG (n=27, 28, 22, 41) | 20.65 (72.42) | 40.06 (74.56) | 4.10 (36.59) | 25.95 (60.73)

8. Secondary Outcome: Increases and Decreases in Lipid Levels
Time Frame: over 24 weeks
Population: Safety Population. All participants having been prescribed at least one dose of study drug.
Measure: Number; unit: participants
Arm/Group | Manic Episode | Hypomanic Episode | Mixed Episode | Depressive Episode
Number analyzed (Participants) | 36 | 31 | 26 | 48
participants
  At Least One Increase for Total Cholesterol (TC) | 18 | 7 | 11 | 20
  At Least One Decrease for TC | 11 | 9 | 10 | 16
  At Least One Increase/Decrease for TC | 19 | 12 | 14 | 26
  Patients Who Increase & Decrease in TC | 10 | 4 | 7 | 10
  ≥1 Increase for High Density Lipoprotein (HDL) | 8 | 5 | 6 | 11
  At Least One Decrease for HDL | 4 | 6 | 5 | 8
  At Least One Increase/Decrease for HDL | 9 | 8 | 7 | 12
  Patients Who Increase & Decrease in HDL | 3 | 3 | 4 | 7
  ≥1 Increase for Low Density Lipoprotein (LDL) | 15 | 8 | 11 | 17
  At Least One Decrease for LDL | 8 | 7 | 7 | 17
  At Least One Increase/Decrease for LDL | 17 | 12 | 12 | 25
  Patients Who Increase & Decrease in LDL | 6 | 3 | 6 | 9
  At Least One Increase for Triglycerides (TG) | 11 | 7 | 6 | 11
  At Least One Decrease for TG | 12 | 7 | 7 | 13
  At Least One Increase/Decrease for TG | 15 | 11 | 8 | 16
  Patients Who Increase & Decrease in TG | 8 | 3 | 5 | 8

9. Secondary Outcome: Mean Change From Baseline to 24 Week Endpoint in Weight
Time Frame: Baseline and 24 weeks
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: kilograms
Arm/Group | Manic Episode | Hypomanic Episode | Mixed Episode | Depressive Episode
Number analyzed (Participants) | 36 | 31 | 26 | 47
kilograms | 1.37 (2.98) | 1.91 (3.44) | 1.78 (4.43) | 2.15 (2.60)

10. Secondary Outcome: Weight Gain Compared to Baseline
Description: Weight gain at anytime more than 7%-15% or 25% of body weight compared to baseline
Time Frame: over 24 weeks
Population: Safety Population. All participants having been prescribed at least one dose of study drug.
Measure: Number; unit: participants
Arm/Group | Manic Episode | Hypomanic Episode | Mixed Episode | Depressive Episode
Number analyzed (Participants) | 36 | 31 | 26 | 48
participants
  No Significant Gain | 30 (2.98) | 26 (3.44) | 18 (4.43) | 42 (2.60)
  >25% | 0 | 0 | 0 | 0
  >15% | 1 | 2 | 1 | 0
  >7% | 5 | 3 | 7 | 5
  Missing Data | 0 | 0 | 0 | 1

11. Secondary Outcome: Wellness Interventional Program for Weight Gain Management in Patients (for Those Who Gain at Anytime More Than 7% of Body Weight, Compared to Baseline)
Time Frame: 24 weeks
Population: Subgroup of patients who gained more than 7% of body weight.
Measure: Number; unit: participants
Groups:
- Weight Gain Subgroup: Patients who gained more than 7% of body weight during the study.
Arm/Group | Weight Gain Subgroup
Number analyzed (Participants) | 24
participants
  Advised to Consult Dietician - No | 8
  Advised to Consult Dietician - Yes | 16
  Performed a Wellness Program - No | 6
  Performed a Wellness Program - Yes | 10
  Number of Wellnes Program Consults - 1 | 5
  Number of Wellnes Program Consults - 2 | 2
  Number of Wellnes Program Consults - 3 | 3
  Patients Losing Weight After Consultation | 8
  Patients Gaining Weight After Consultation | 8
  Patients with Stable Weight After Consultation | 0

12. Secondary Outcome: MATHYS Total Score at Baseline - According to Thymic Reactivity Assessment
Description: A visual analogic scale consisting of 20 items. Items scores vary from 0 (inhibition of the state evaluated by the item) to 10 (excitation for the evaluated state), except for items 5 to 10 and 17 and 18, which are inversed and are consequently to be reversed before the analysis. Total score is sum of the 20 items and can vary from 0 to 200.
Time Frame: Baseline
Population: Intention to treat. Number of participants with baseline and at least one non-missing postbaseline value.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Thymic Hypo-Reactive; Thymic Hyper-Reactivity; Neither: As assessed by the investigator according to his clinical experience.
Arm/Group | Thymic Hypo-Reactive | Thymic Hyper-Reactivity | Neither
Number analyzed (Participants) | 30 | 101 | 10
units on a scale | 81.24 (30.81) | 122.49 (32.01) | 117.26 (26.41)

13. Secondary Outcome: Change From Baseline to 6 Week and 24 Week Endpoints in HAMA Total Scores - According to Thymic Reactivity Assessment
Description: as for outcome 3
Time Frame: Baseline, 6 Weeks, 24 Weeks
Population: Intention to treat. Number of participants with baseline and at least one non-missing postbaseline value.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Thymic Hypo-Reactivity; Thymic Hyper-Reactivity; Neither: As assessed by the investigator according to his clinical experience.
Arm/Group | Thymic Hypo-Reactivity | Thymic Hyper-Reactivity | Neither
Number analyzed (Participants) | 30 | 101 | 10
units on a scale
  Baseline (n=30, 101, 10) | 12.87 (7.09) | 12.63 (7.95) | 11.40 (7.95)
  Change from 6 Week Endpoint (n=29, 93, 10) | -4.93 (5.62) | -5.96 (6.56) | -4.30 (3.95)
  Change from 24 Week Endpoint (n=30, 99, 10) | -4.83 (5.94) | -5.65 (7.39) | -6.90 (7.43)

14. Secondary Outcome: Change From Baseline to 6 Week and 24 Week Endpoints in HAMD-17 Total Scores - According to Thymic Reactivity Assessment
Description: as for outcome 2
Time Frame: Baseline, 6 Weeks, 24 Weeks
Population: Intention to treat. Number of participants with baseline and at least one non-missing postbaseline value.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Thymic Hypo-Reactivity | Thymic Hyper-Reactivity | Neither
Number analyzed (Participants) | 30 | 101 | 10
units on a scale
  Baseline (n=29, 100, 10) | 14.48 (7.02) | 10.64 (6.85) | 9.50 (7.01)
  Change from 6 Week Endpoint (n=28, 90, 10) | -6.61 (5.02) | -4.89 (6.62) | -4.00 (5.12)
  Change from 24 Week Endpoint (n=28, 98, 10) | -6.48 (4.32) | -4.55 (7.58) | -3.80 (4.85)

15. Secondary Outcome: Change From Baseline to 6 Week and 24 Week Endpoints in YMRS Total Scores - According to Thymic Reactivity Assessment
Description: as for outcome 4
Time Frame: Baseline, 6 Weeks, 24 Weeks
Population: Intention to treat. Number of participants with baseline and at least one non-missing postbaseline value.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Thymic Hypo-Reactivity | Thymic Hyper-Reactivity | Neither
Number analyzed (Participants) | 30 | 101 | 10
units on a scale
  Baseline (n=27, 101, 10) | 4.48 (7.99) | 16.50 (10.65) | 10.00 (7.24)
  Change from 6 Week Endpoint (n=26, 93, 10) | -2.38 (7.90) | -10.45 (8.46) | -6.50 (4.70)
  Change from 24 Week Endpoint (n=27, 99, 10) | -1.70 (5.19) | -11.29 (9.89) | -7.60 (5.52)

16. Secondary Outcome: Emotional Reactivity With the Physiological Measure of Heart Rate
Description: to assess emotional reactivity with the physiological measure of heart rate, recorded as a function of slides sessions from the International Affective Picture System, in a defined subgroup of patients
Time Frame: 12 weeks
Population: Measures were to be collected at only one site. Not enough data to analyze.
Measure: Mean (Standard Deviation); unit: beats per minute
Arm/Group | Manic Episode | Hypomanic Episode | Mixed Episode | Depressive Episode
Number analyzed (Participants) | 0 | 0 | 0 | 0

17. Secondary Outcome: Emotional Reactivity With the Physiological Measure of Skin Conductance
Description: To assess emotional reactivity with the physiological measure of skin conductance, recorded as a function of slides sessions from the International Affective Picture System, in a defined subgroup of patients.
Time Frame: 12 weeks
Population: Measures were to be collected at only one site. Not enough data to analyze.
Measure: Mean (Standard Deviation); unit: microvolts
Arm/Group | Manic Episode | Hypomanic Episode | Mixed Episode | Depressive Episode
Number analyzed (Participants) | 0 | 0 | 0 | 0

18. Secondary Outcome: Emotional Reactivity With the Physiological Measure of Startle Reflex Response - Latency of Blink
Description: To assess emotional reactivity with the physiological measure of startle reflex response by measuring the latency of the blink, recorded as a function of slides sessions from the International Affective Picture System, in a defined subgroup of patients.
Time Frame: 12 weeks
Population: Measures were to be collected at only one site. Not enough data to analyze.
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Manic Episode | Hypomanic Episode | Mixed Episode | Depressive Episode
Number analyzed (Participants) | 0 | 0 | 0 | 0

19. Secondary Outcome: Emotional Reactivity With the Physiological Measure of Startle Reflex Response - Amplitude of Blink
Description: To assess emotional reactivity with the physiological measure of startle reflex response - by measuring the amplitude of the blink, recorded as a function of slides sessions from the International Affective Picture System, in a defined subgroup of patients.
Time Frame: 12 weeks
Population: Measures were to be collected at only one site. Not enough data to analyze.
Measure: Mean (Standard Deviation); unit: microvolts
Arm/Group | Manic Episode | Hypomanic Episode | Mixed Episode | Depressive Episode
Number analyzed (Participants) | 0 | 0 | 0 | 0

20. Primary Outcome: Baseline MATHYS Assessment - Principal Component Analysis and Orthogonal Transformation Matrix
Description: This analysis indicates whether the total score is correct and provides enough information, or if subscores need to be calculated. Eigen value, proportion and cumulative are statistical parameters from the Principal Component Analysis, given for each factor.
Time Frame: Baseline
Population: Matrix based on data from all 141 participants.
Measure: Number; unit: value
Arm/Group | Eigen Value | Proportion | Cumulative
Number analyzed (Participants) | 141 | 141 | 141
value
  Factor 1 | 8.77 | 0.4383 | 0.4383
  Factor 2 | 2.01 | 0.1006 | 0.5389
  Factor 3 | 1.19 | 0.0594 | 0.5984
  Factor 4 | 1.042 | 0.0521 | 0.6505
  Factor 5 | 0.98 | 0.0490 | 0.6995
  Factor 6 | 0.79 | 0.0397 | 0.7392
  Factor 7 | 0.69 | 0.0347 | 0.7739
  Factor 8 | 0.64 | 0.0322 | 0.8061
  Factor 9 | 0.56 | 0.0280 | 0.8341
  Factor 10 | 0.54 | 0.0268 | 0.8608
  Factor 11 | 0.45 | 0.0227 | 0.8836
  Factor 12 | 0.44 | 0.0219 | 0.9055
  Factor 13 | 0.37 | 0.0186 | 0.9241
  Factor 14 | 0.34 | 0.0171 | 0.9412
  Factor 15 | 0.28 | 0.0139 | 0.9551
  Factor 16 | 0.26 | 0.0131 | 0.9682
  Factor 17 | 0.20 | 0.0100 | 0.9782
  Factor 18 | 0.18 | 0.0091 | 0.9873
  Factor 19 | 0.14 | 0.0071 | 0.9944
  Factor 20 | 0.11 | 0.0056 | 1.0000

ADVERSE EVENTS:
Arm/Group | Olanzapine
Serious Adverse Events (participants affected / at risk) | 14
Other Adverse Events (participants affected / at risk) | 53
SERIOUS ADVERSE EVENTS; cells are participants affected / at risk (number of events):
Term (organ system) | Olanzapine
Gastric ulcer (Gastrointestinal disorders) | 1/141 (1)
Cholecystitis (Hepatobiliary disorders) | 1/141 (1)
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1/141 (1)
Alcoholism (Psychiatric disorders) | 1/141 (1)
Anxiety (Psychiatric disorders) | 1/141 (1)
Bipolar I disorder (Psychiatric disorders) | 5/141 (5)
Depression (Psychiatric disorders) | 4/141 (4)
Suicide attempt (Psychiatric disorders) | 1/141 (1)
Arteritis (Vascular disorders) | 1/141 (2)
OTHER ADVERSE EVENTS; cells are participants affected / at risk (number of events):
Term (organ system) | Olanzapine
Palpitations (Cardiac disorders) | 1/141 (1)
Vertigo (Ear and labyrinth disorders) | 1/141 (1)
Hyperprolactinaemia (Endocrine disorders) | 1/141 (1)
Hypothyroidism (Endocrine disorders) | 1/141 (1)
Eye pruritus (Eye disorders) | 1/141 (1)
Vision blurred (Eye disorders) | 2/141 (2)
Visual disturbance (Eye disorders) | 1/141 (1)
Abdominal pain (Gastrointestinal disorders) | 1/141 (1)
Constipation (Gastrointestinal disorders) | 7/141 (7)
Diarrhoea (Gastrointestinal disorders) | 2/141 (3)
Dry mouth (Gastrointestinal disorders) | 8/141 (8)
Gastrointestinal disorder (Gastrointestinal disorders) | 1/141 (1)
Nausea (Gastrointestinal disorders) | 1/141 (1)
Salivary hypersecretion (Gastrointestinal disorders) | 1/141 (1)
Vomiting (Gastrointestinal disorders) | 2/141 (2)
Asthenia (General disorders) | 3/141 (3)
Food allergy (Immune system disorders) | 1/141 (1)
Bronchitis (Infections and infestations) | 1/141 (1)
Influenza (Infections and infestations) | 1/141 (1)
Alanine aminotransferase increased (Investigations) | 1/141 (1)
Blood creatine phosphokinase increased (Investigations) | 1/141 (1)
Blood triglycerides increased (Investigations) | 1/141 (1)
Gamma-glutamyltransferase increased (Investigations) | 2/141 (2)
Red blood cell sedimentation rate increased (Investigations) | 1/141 (1)
Transaminases increased (Investigations) | 1/141 (1)
Weight increased (Investigations) | 3/141 (3)
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 1/141 (1)
Increased appetite (Metabolism and nutrition disorders) | 2/141 (2)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1/141 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 1/141 (1)
Akathisia (Nervous system disorders) | 1/141 (1)
Cognitive disorder (Nervous system disorders) | 1/141 (1)
Dizziness (Nervous system disorders) | 2/141 (2)
Dysarthria (Nervous system disorders) | 1/141 (1)
Headache (Nervous system disorders) | 1/141 (1)
Hypertonia (Nervous system disorders) | 1/141 (1)
Paraesthesia (Nervous system disorders) | 1/141 (1)
Restless legs syndrome (Nervous system disorders) | 1/141 (1)
Sedation (Nervous system disorders) | 1/141 (1)
Somnolence (Nervous system disorders) | 7/141 (8)
Tremor (Nervous system disorders) | 7/141 (7)
Agitation (Psychiatric disorders) | 1/141 (1)
Depression (Psychiatric disorders) | 1/141 (1)
Loss of libido (Psychiatric disorders) | 2/141 (2)
Memory impairment (Psychiatric disorders) | 1/141 (1)
Sleep disorder (Psychiatric disorders) | 1/141 (1)
Suicidal ideation (Psychiatric disorders) | 2/141 (2)
Suicide attempt (Psychiatric disorders) | 1/141 (1)
Urinary tract disorder (Renal and urinary disorders) | 1/141 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1/141 (1)
Photosensitivity reaction (Skin and subcutaneous tissue disorders) | 1/141 (1)
Arteritis (Vascular disorders) | 1/141 (2)

LIMITATIONS AND CAVEATS:
Fewer patients than planned were enrolled in the study. Not all the analyses (Principal Component Analysis, scree plot to define the structure) could be provided due to the specific formatting of the clinicaltrials.gov databank.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days